CLINICAL TRIAL: NCT00334087
Title: Assessment of Pregnancy History, Birth Outcome, Feeding and Oral Practices With Development of Early Childhood Caries in Offspring of Women Who Have Not Participated in Previous Birth Preparation Class
Brief Title: The Relation Between Pregnancy,Birth Outcome, Feeding , Oral Hygiene Habits and Early Childhood Caries Development.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: boquita HMO-CTIL
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Dental Caries
Keywords: primary dental prevention; early childhood caries; prenatal oral care
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: feeding habits

SUMMARY:
* 200 children between ages 36 to 48 months will be invited for a regular dental examination
* Parameters to be investigated

  1. Pregnancy history
  2. Birth outcome
  3. Child's general health
  4. Feeding habits
  5. Oral hygiene habits
  6. Dmft caries index
  7. Congenital enamel defects

DETAILED DESCRIPTION:
Severe Early Childhood Caries is a condition whereby very young children suffer multiple caries. The value of a pre- perinatal preventive approach is currently being examined in the dental literature. At Hadassah, a Pilot Study is currently underway to test the feasibility of a comprehensive Baby Clinic designed to prevent Severe Early Childhood Caries. The pilot study in cooperation with the Woman's Health Center and with the midwives and the breastfeeding counselors of the maternity unit. Lectures are given by pediatric dentists to parents of firstborn children attending Hadassah's Birth Preparation Class, emphasis is given to the importance of breastfeeding and other feeding habits in the emotional, physical, nutritional and immunological development of the future baby. In addition the effect of these feeding habits on the dental/oral aspects, relevant for the developing dentition.

After birth the parents are invited to come with their babies around 12 months for the first dental examination and follow up according to individual risk for caries development. The current proposed study will be a control group from offspring of women who have participated previous Sessions Hadassah's Birth Preparation Class ("Historical Controls" before the Baby Clinic project)

ELIGIBILITY:
Inclusion Criteria:

* children born in previous Sessions Hadassah's Birth Preparation Class " before the Baby Clinic project)

Exclusion Criteria:

* children not born in previous Sessions Hadassah's Birth Preparation Class " before the Baby Clinic project)

Ages: 36 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Mamber, DMD, Principal Investigator — Hadassah Medical Organization IRB
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Gomez SS, Weber AA. Effectiveness of a caries preventive program in pregnant women and new mothers on their offspring. Int J Paediatr Dent. 2001 Mar;11(2):117-22. doi: 10.1046/j.1365-263x.2001.00255.x. PMID 11310134